CLINICAL TRIAL: NCT05586685
Title: Effect of Diaphragmatic Release on Upper Crossed Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Mohamed Abd El-Rahem, teaching assistant at basic science department, faculty of physical therapy egyptian chinese university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.tREC/012/003917
Record Dates: First submitted 2022-10-15; First posted 2022-10-19 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Neck Muscle Issue; Kyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the patients and investigator do not know the groups receive treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GroupA diaphragmatic release + conventional (Experimental): Group A: diaphragmatic release +conventional The patients will be positioned in the supine position. The therapist stood at the head of the patient contact thoracic cage and ask the patient to take inspiration and move laterally then ask the patient to expire.
  conventional Subjects will form the letter 'Y' with their arms then they will flex their elbows and move into a position of shoulder extension so that their arms will form the letter 'w L to Y Exercise: Subjects will begin with arms abducted to 90° and elbows flexed to 90° Chin tucks: Subjects will length the neck by pushing the chin into the table in an entirely posterior motion stretch the pectoral area from the supine lying position
  Interventions: Other: effect of diaphragmatic release on upper crossed syndrome
- Group B: conventional (Experimental): Group B: conventional posture correction exercises Subjects will form the letter 'Y' with their arms then they will flex their elbows and move into a position of shoulder extension, so that their arms will form the letter 'w L to Y Exercise: Subjects will begin with arms abducted to 90° and elbows flexed to 90° Chin tucks : Subjects will length the neck by pushing the chin into the table in an entirely posterior motion stretch pectoral area from supine lying position
  Interventions: Other: effect of diaphragmatic release on upper crossed syndrome

INTERVENTIONS:
Other: effect of diaphragmatic release on upper crossed syndrome — The patients will be positioned in the supine position. The therapist stood at the head of the patient.therapist make manual contact of ribs and ask patient to inspire the move ribs laterally and then expire
  conventional exercise Subjects will form the letter 'Y' with their arms then they will flex their elbows and move into a position of shoulder extension, so that their arms will form the letter 'w L to Y Exercise: Subjects will begin with arms abducted to 90° and elbows flexed to 90° Chin tucks : Subjects will length the neck by pushing the chin into the table in an entirely posterior motion stretch pectoral area from supine lying position

SUMMARY:
the study aims to investigate the effectiveness of diaphragmatic release on upper crossed syndrome

DETAILED DESCRIPTION:
Poor posture typically causes upper cross syndrome, resulting in neck pain. Neck pain is the most common reason for patients to visit healthcare professionals. This syndrome can cause dysfunctional tone in posture and muscular disparity of the head, neck, and shoulder region . Evidence suggests that 6-48% of the upper crossed syndrome population complain of pain in the shoulder girdle and cervicothoracic region.

Many disorders are linked with the upper crossed syndrome, including migraine headaches; chronic headaches; Subacromial impingement; biceps tendinitis; thoracic outlet syndrome; degeneration of the cervical spine; and joint dysfunction at the C1-C2 segment, C4-C5 segment, cervicothoracic joint, and T4-T5 segment.

Upon the available research studies, there is no study conducted to investigate the effect of diaphragmatic release on upper crossed syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 17 to 22 years .
* Body Mass Index from 20 to 25 kg/m².
* All participants have an intensity of neck pain on VAS (4-8) (moderate cases).
* The subjects were chosen from both sexes.
* All participants have kyphosis angle ≥42°
* All participants have mechanical neck pain and FHP (craniovertebral angle CVA < 49).

Exclusion Criteria:

* Malignancy
* Fractures of the cervical spine
* Cervical radiculopathy or myelopathy
* Vascular syndromes such as vertebrobasilar insufficiency
* Rheumatoid arthritis
* Neck or upper back surgery
* Taking anticoagulants
* Local infection
* Whiplash injury

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
chest expansion with tape measurement | up to four weeks
  using tape to measure chest expansion during inspiration and expiration at axillary level and at the level of T10

SECONDARY OUTCOMES:
pain intensity with pain numerical scale scale | up to four weeks
  The subject was instructed to place a vertical mark on the line to indicate his/her pain which zero is no pain and ten being severe pain.